CLINICAL TRIAL: NCT05837117
Title: Sexual Dysfunction in Palliative Care Patients: An Assessment of Patient's Perspective
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0495; NCI-2022-10774 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient's Perspective: Participants will complete a questionnaire about sexual wellbeing, sexual dysfunction, and communication with your provider on this topic. Participants may choose to complete the questionnaire electronically (via email link), in-person, or over the phone, whichever you prefer. Your demographic information (such as age, gender, ethnicity, marital status, and cancer diagnosis) will be collected from your medical record. Some of this information may also be asked of you during the questionnaire.
  Interventions: Behavioral: Patient's Perspective

INTERVENTIONS:
Behavioral: Patient's Perspective — Participants will complete a questionnaire about sexual wellbeing, sexual dysfunction, and communication with your provider on this topic.
  Participants/Researchers will learn about your attitudes, beliefs, and feelings about sexual well-being

SUMMARY:
To learn about the communications that Supportive Care patients receive about sexual well-being from their healthcare provider. Researchers also want to learn about your attitudes, beliefs, and feelings about sexual well-being.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the frequency of discussion about sexual dysfunction in palliative care patients.
2. To evaluate the impact of cancer diagnosis and treatment on patient's sexual life.

Secondary Objectives:

1. To evaluate patient self-reported severity of sexual dysfunction
2. To evaluate the proportion of patients suffering distress from body image concerns
3. To identify patient self-reported barriers that prevent discussion about sexual dysfunction
4. To evaluate patient self-reported impact of sexual dysfunction on their wellbeing

ELIGIBILITY:
Inclusion Criteria:

* All patients who are evaluated as follow-ups in the Supportive Care clinic, and able to voluntarily consent to participate in the study
* Patients must be able to understand, read, write, and speak English
* Diagnosis of cancer
* Patients who are 18 years of age or older

Exclusion criteria:

* New patients (consults)
* Patient who have declined to participate, or who are unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaires | through study completion an average of year

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bramati, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org